CLINICAL TRIAL: NCT04753970
Title: Retinal Vasoreactivity is a Marker for Cerebral Small Vessel Disease Progression
Brief Title: Retina is a Marker for Cerebrovascular Heath
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michelle P. Lin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-000087
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Small Vessel Diseases; Cerebral Autosomal Dominant Arteriopathy With Subcortical Infarcts and Leukoencephalopathy; Cerebral Microbleeding; Sporadic White Matter Disease
MeSH Terms: conditions — Cerebral Small Vessel Diseases; CADASIL | interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cilostazol (Experimental): Cilostazol 100mg BID
  Interventions: Drug: Cilostazol
- No intervention (No Intervention)

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 100mg BID
  Arms: Cilostazol

SUMMARY:
Cerebral small vessel disease (SVD), present in 80-94% of adults over age 65 years, increases the risk of stroke by 2-fold, and dementia by 2.3-fold. There is currently no treatment to slow SVD progression. This study aims to test whether impaired cerebral and retinal vasoreactivity may serve as biomarker for SVD progression, and to evaluate the safety and efficacy of cilostazol (antiplatelet agent with vasodilatory and anti-inflammatory properties) for the treatment of SVD.

DETAILED DESCRIPTION:
This is a prospective, observational nested pilot randomized controlled study to discover retinal biomarkers that would predict cerebral small vessel disease progression, and evaluate the safety/efficacy of cilostazols in slowing SVD progression. Twenty CADASIL, 40 sWMD, 20 lobar CMB, and 20 age-matched healthy controls from the Mayo Clinic Florida Familial Cerebrovascular Disease Registry and neurology clinic will be recruited. All participants will undergo OCTA retinal scan, MRI-BOLD brain scan, cognitive battery evaluation, and blood sample at baseline and a 12-month follow-up visit. Key outcome measures are: RVR, CVR, cognition, WMH volume, and CMB volume. The 40 patients diagnosed in the course of routine clinical care with sWMD will be randomized in 1:1 ratio to receive cilostazol 100mg bid (or 50 mg bid if taking medications known to affect metabolism of cilostazol) or no cilostazol, and followed for WMD progression, and secondarily for changes in cognition, RVR and CVR. Flow diagram below outlines the study design. Note that in addition to what is shown in the trial flow diagram, patients will have telephone visits between baseline and 12 month clinic visits biweekly for 3 months and then monthly thereafter. These visits will consist of a survey for adverse events and at the 1-, 3-, 6- and 9-month telephone visits patients will also get a modified Rankin scale assessment, a Six-item screener (cognitive assessment) and a PHQ-2 (depression screen).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 yo.
* Diagnosis of CADASIL, sporadic WMD or lobar CMB and age-matched healthy controls (eg. patient's spouse or unrelated friends without SVD)

Exclusion Criteria:

* Age<18yo
* Pregnant
* Breast feeding
* Unable to follow commands
* Unable to tolerate MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
white matter disease volume | 1 year
  change in total white matter disease volume

SECONDARY OUTCOMES:
cognition | 1 year
  global Z-score and by cognitive domain
stroke | 1 year
  ischemic stroke or hemorrhagic stroke
cerebrovasoreactivity | 1 year
  change in blood oxygen level dependence (BOLD) per unit of end tidal PCO2 mmHg
retinal vasoreactivity | 1 year
  change in retinal vessel density pre/post CO2 challenge

CONTACTS AND LOCATIONS:
Overall Officials: Michelle P Lin, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No